CLINICAL TRIAL: NCT06867718
Title: A Phase 2 Study of Once-Daily RGT001-075 Compared With Placebo in Participants Who Have Obesity or Are Overweight With Weight-Related Comorbidities (COMO-1)
Brief Title: Study of Once-Daily Oral RGT001-075 Compared With Placebo in Adults With Obesity or Are Overweight With Weight-Related Health Conditions
Acronym: COMO-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regor Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGT001-075-205
Record Dates: First submitted 2025-02-14; First posted 2025-03-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obesity or Overweight
Keywords: GLP-1 receptor agonist (GLP-1 RA); Obesity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- RGT1 (Experimental): Study Drug: RGT001-075 (Dose 1)
  Interventions: Drug: RGT001-075
- RGT2 (Experimental): Study Drug: RGT001-075 (Dose 2)
  Interventions: Drug: RGT001-075
- RGT3 (Experimental): Study Drug: RGT001-075 (Dose 3)
  Interventions: Drug: RGT001-075
- RGT4 (Experimental): Study Drug: RGT001-075 (Dose 4)
  Interventions: Drug: RGT001-075
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: RGT001-075 — RGT001-075 is a small molecule GLP-1 agonist
  Arms: RGT1; RGT2; RGT3; RGT4
Drug: Placebo Comparator — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a phase 2, 36-week randomized, double-blind, placebo-controlled, parallel arm study that will evaluate the safety, tolerability, weight loss efficacy, pharmacodynamic effects, and pharmacokinetics of RGT001-075 in adults who are obese (BMI ≥30 kg/m²) or who are overweight (BMI ≥27 kg/m²) with at least one weight-related comorbidity. RGT001-075 or matching placebo will be administered once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-75 years (inclusive) at the time of signing informed consent.
2. Hemoglobin A1c (HbA1c) <6.5% at screening.
3. BMI ≥30 kg/m².
4. BMI ≥27 kg/m² and <30 kg/m² with at least 1 weight-related comorbidity:

   * hypertension
   * dyslipidemia
   * cardiovascular (CV) disease
   * obstructive sleep apnea
5. Have a stable body weight (< 5% change) for the 3 months prior to randomization.

Exclusion Criteria (Obesity Related):

1. Have obesity induced by other endocrine disorders (for example, Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome).
2. Have a prior or planned surgical treatment for obesity.
3. Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months before screening such as mucosal ablation, gastric artery embolization, intragastric balloon, duodenal-jejunal endoluminal liner.
4. Have been treated with prescribed or OTC drugs or alternative remedies that promote weight loss within the last 3 months before screening.

Exclusion Criteria (Medical Conditions)

1. Diabetes.
2. Have a history of acute or chronic pancreatitis.
3. Have current symptomatic gallbladder disease or biliary disease.
4. Have known liver disease other than MASLD.
5. Have a known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or medullary thyroid carcinoma (MTC).
6. Have a serum calcitonin ≥20 pg/mL.
7. Have an eGFR <30 mL/min/1.73 m², as determined by the central laboratory at screening.
8. Have a history of Major Depressive Disorder (MDD) or other severe psychiatric disorders (e.g., schizophrenia or bipolar disorder) within the last 2 years.
9. Have had any exposure to GLP-1 analogs, or other related compounds within the prior 3 months or any prior history of clinically significant side effects from GLP-1 receptor agonist (GLP-1 RA) or other related compounds containing GLP-1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight at Week 36 | Baseline and 36 weeks
  Least Squares (LS) mean using mixed model repeated measures (MMRM)

SECONDARY OUTCOMES:
Percent change from baseline in body weight at Week 26 | Baseline and 26 weeks
  Least Squares (LS) mean using mixed model repeated measures (MMRM)
Incidence of treatment emergent adverse events (TEAEs), TESAEs, TEAESIs overall | Baseline through week 36
  To evaluate the safety and tolerability of RGT001-075 for weight loss in adults who are obese, or overweight with at least one weight-related comorbidity
Ambulatory Blood Pressure Monitoring (ABPM) | Baseline, 26 weeks
  The ABPM device will be attached to the nondominant arm, and participants will be instructed to wear the monitor for a 24- to 27-hour period.
AUC0-last | week 15
  Area under the serum concentration curve from time-zero to the last quantifiable concentration of RGT001-075
AUC0-inf | week 15
  Area under curve from time zero to time infinite
Cmax | week15
  Maximum concentration of RT001-075
Tmax | week 15
  Time to achieve maximum concentration of RT001-075
t1/2 | week 15
  Terminal half-life of RGT001-075

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Synexus Clinical Research, Phoenix, Arizona
  - Velocity Clinical Research, Huntington Park, California
  - Angels Clinical Research, Doral, Florida
  - Optimal Research, Melbourne, Florida
  - Angels Clinical Research, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Synexus Clinical Research, The Villages, Florida
  - Javara-Privia Medical Group, Georgia LLC, Savannah, Georgia
  - Javara-Privia Medical Group, Georgia, LLC, Thomasville, Georgia
  - Synexus Clinical Research, Evansville, Indiana
  - Velocity Clinical Research, Valparaiso, Indiana
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Velocity Clinical Research, Baton Rouge, Louisiana
  - Velocity Clinical Research, Rockville, Maryland
  - Mankato Clinic-East Main Street-Javara, Mankato, Minnesota
  - Synexus Clinical Research, Richfield, Minnesota
  - Synexus Clinical Research, Creve Coeur, Missouri
  - Velocity Clinical Research, Omaha, Nebraska
  - Premier Health Research-Sparta-Objective Health, Sparta, New Jersey
  - Velocity Clinical Research, Vestal, New York
  - Javara-Tryon Medical Partners, PLLC, Charlotte, North Carolina
  - Velocity Clinical Research, Durham, North Carolina
  - Velocity Clinical Research, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Velocity Clinical Research, East Greenwich, Rhode Island
  - Velocity Clinical Research, Dallas, Texas
  - Synexus Clinical Research, Dallas, Texas
  - Synexus Clinical Research, San Antonio, Texas
  - Javara-Privia Medical Group Gulf Coast PLLC, The Woodlands, Texas
  - Velocity Clinical Research, Waco, Texas
  - Synexus Clinical Research, Salt Lake City, Utah
  - Velocity Clinical Research, West Jordan, Utah
  - Velocity Clinical Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor recognizes that sharing anonymized data and other information from clinical trials can enhance biomedical research. The Sponsor is following ongoing discussions among industry, academia, and other stakeholders regarding data sharing. Industry and academic partners hold various positions on the amount, types, and forms of data that will be useful l to the research community, the public, and the process for sharing. As a small, young company, the Sponsor awaits further guidance and input from industry participants on best practices before issuing a comprehensive data sharing plan. For now, Sponsor defers a description of what data will be shared and the process for doing so.